CLINICAL TRIAL: NCT06426810
Title: A Prospective Randomized Study Comparing Electrosurgical Bipolar Systems Versus Conventional Electrocautery After Sentinel Lymph Node Biopsy in Obese or Preoperative Chemotherapy Treated Breast Cancer Patients
Brief Title: Electrosurgical Bipolar Systems Versus Conventional Electrocautery After SLNBx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jong-Ho Cheun, Clinical Professor, SMG-SNU Boramae Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-2024-18
Record Dates: First submitted 2024-05-07; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrosurgical bipolar systems group (Experimental): Study participants using a electrosurgical bipolar energy system will undergo sentinel lymph node biopsy using only LigaSure during the surgery.
  Interventions: Device: Electrosurgical bipolar system (LigaSure)
- Conventional electrocautery group (No Intervention): Study participants using a conventional electrocautery will undergo sentinel lymph node biopsy using conventional bovie electrocautery during the surgery.

INTERVENTIONS:
Device: Electrosurgical bipolar system (LigaSure) — Study participants using a electrosurgical bipolar energy system will undergo sentinel lymph node biopsy using only LigaSure during the surgery.
  Arms: Electrosurgical bipolar systems group

SUMMARY:
The efficacy of electrosurgical bipolar systems in axillary lymph node dissection for breast cancer surgery is well known. In this study, the investigators aim to determine whether using electrosurgical bipolar systems helps reduce seroma formation in high-risk patients undergoing sentinel lymph node biopsy (SLNB) for breast cancer surgery. The investigators will focus on patients who are expected to experience high drainage output after SLNB, especially those who are obese (BMI>25) or have undergone preoperative chemotherapy.

DETAILED DESCRIPTION:
The most common complications of breast cancer surgery are lymphorrhea and seroma. Seroma increases the length of hospital stay, the duration of outpatient treatment, and patient discomfort. Persistent seroma can lead to re-hospitalization due to wound infection caused by repeated aspirations. Seroma generally occurs in 10% to 85% of cases after breast cancer surgery. Risk factors associated with seroma or lymphorrhea identified in previous studies include age over 60, high BMI, tumor size, preoperative chemotherapy, extent of breast tissue resection, number of lymph nodes removed, and number of lymph node metastases.

Efforts to reduce seroma after breast cancer surgery include meticulous techniques such as sharp dissection, the use of monopolar energy devices, and ligation of blood vessels and lymphatics. Recently, the bipolar energy sealing system has been increasingly used. LigaSure, which uses electric energy and pressure to denature collagen and elastin in tissue, has been shown to reduce surgical time and medical costs compared to traditional clamp-and-tie methods and advanced sealing systems in various surgeries, including breast cancer.

In breast cancer surgery, using a electrosurgical bipolar systems for ligating blood vessels and lymph nodes has several potential advantages. Traditional ligation using sutures or monopolar energy devices can be influenced by surgical technique and has drawbacks such as thermal injury to surrounding tissue. In contrast, the bipolar energy sealer applies both electric energy and pressure simultaneously, minimizing thermal injury to surrounding tissue while ensuring permanent vessel and lymphatic ligation.

A 2008 prospective study showed that using bipolar energy sealers in axillary dissection allowed for earlier removal of drains compared to conventional methods. Other studies have shown less blood loss, lower drainage output, and shorter hospital stays during surgery. Recent research has also reported new applications of bipolar energy sealers in skin-sparing mastectomy, indicating active use in breast surgery overseas. A study conducted at Severance Hospital in South Korea found that using bipolar energy sealers reduced drainage.

However, most of these studies were conducted abroad with a small number of reported cases, and the results mainly concern axillary lymph node dissection (ALND), which is where seroma is most often formed. With the decreasing trend of ALND due to advances in preoperative chemotherapy and radiotherapy, there is a lack of studies on whether using electrosurgical bipolar systems helps reduce seroma formation after sentinel lymph node biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20-80
* Candidates for breast-conserving surgery and axillary sentinel lymph node biopsy
* BMI over 25 or those who have received preoperative chemotherapy
* Overall performance status of Eastern Cooperative Oncology Group (ECOG) 0-2
* Participants who understand the study contents and can provide written consent
* Participants without evidence of distant metastasis

Exclusion Criteria:

* Those with suspected axillary lymph node enlargement or metastasis on preoperative imaging (breast MRI, chest CT, breast ultrasound)
* Among patients who had confirmed lymph node metastasis before neoadjuvant chemotherapy, whose preopreative image showed residual disease at axillary lymph node
* Those planning for mastectomy
* Those planning for axillary lymph node dissection without SLNBx
* Male breast cancer patients
* Patients with bilateral breast cancer
* Illiterate individuals, foreigners, or others who cannot read or understand the consent form
* Individuals who voluntarily decide not to participate in the study or do not sign the consent form
* Those judged by the researcher to be inappropriate for participation in this study
* Study participants who did not have a drain inserted in the surgical area
* If the randomized device is not used due to surgical room conditions (e.g., unavailability due to other emergency surgeries, device malfunction) and another device is substituted

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2027-04-07 (Estimated); Study Completion 2027-04-07 (Estimated)

PRIMARY OUTCOMES:
Drainage amount | Up to four weeks
  Total drainage amount from axilla after surgery (ml)

SECONDARY OUTCOMES:
Drainage amount during admission | Up to one week
  Total drainage amount from axilla before discharge (ml)
Operation time | Up to 2 hours
  Operation time during axillar surgery (min)
Complication | At one month of surgery
  Complications of axilla
Draine removal days | Up to two weeks
  Days before drain removal (days)

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Ho Cheun, M.S., Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- SMG-SNU Boramae medical center, Seoul, Dongjak-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Bemmel AJ, van de Velde CJ, Schmitz RF, Liefers GJ. Prevention of seroma formation after axillary dissection in breast cancer: a systematic review. Eur J Surg Oncol. 2011 Oct;37(10):829-35. doi: 10.1016/j.ejso.2011.04.012. Epub 2011 Aug 17. PMID 21849243
- [Background] Manouras A, Markogiannakis H, Genetzakis M, Filippakis GM, Lagoudianakis EE, Kafiri G, Filis K, Zografos GC. Modified radical mastectomy with axillary dissection using the electrothermal bipolar vessel sealing system. Arch Surg. 2008 Jun;143(6):575-80; discussion 581. doi: 10.1001/archsurg.143.6.575. PMID 18559751
- [Background] Nespoli L, Antolini L, Stucchi C, Nespoli A, Valsecchi MG, Gianotti L. Axillary lymphadenectomy for breast cancer. A randomized controlled trial comparing a bipolar vessel sealing system to the conventional technique. Breast. 2012 Dec;21(6):739-45. doi: 10.1016/j.breast.2012.08.003. Epub 2012 Sep 7. PMID 22959311
- [Background] Cortadellas T, Cordoba O, Espinosa-Bravo M, Mendoza-Santin C, Rodriguez-Fernandez J, Esgueva A, Alvarez-Vinuesa M, Rubio IT, Xercavins J. Electrothermal bipolar vessel sealing system in axillary dissection: a prospective randomized clinical study. Int J Surg. 2011;9(8):636-40. doi: 10.1016/j.ijsu.2011.08.002. Epub 2011 Sep 10. PMID 21925293
- [Background] Miyagi K, Rossi SH, Malata CM, Forouhi P. Novel use of LigaSure Impact electrosurgical bipolar vessel sealing system in skin-sparing mastectomy. J Plast Reconstr Aesthet Surg. 2015 Jun;68(6):e126-8. doi: 10.1016/j.bjps.2015.01.005. Epub 2015 Jan 26. No abstract available. PMID 25682592
- [Background] Park HS, Lee J, Kim JY, Park JM, Kwon Y. A Prospective Randomized Study to Compare Postoperative Drainage After Mastectomy Using Electrosurgical Bipolar Systems and Conventional Electro-Cautery. J Breast Cancer. 2022 Aug;25(4):307-317. doi: 10.4048/jbc.2022.25.e29. Epub 2022 Jun 27. PMID 35914746

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT06426810/Prot_SAP_000.pdf